CLINICAL TRIAL: NCT05993468
Title: A Mixed-Methods Pilot Study of a Trauma-Sensitive Mindfulness and Compassion Intervention
Brief Title: A Pilot Study of a Trauma-Sensitive Mindfulness and Compassion Intervention
Status: Completed | Type: Observational
Sponsor: Modum Bad (Other)
Responsible Party: Principal Investigator, KAVrabel, Research director, Modum Bad
Other Study IDs: Trauma Outpatient Unit
Record Dates: First submitted 2023-06-26; First posted 2023-08-15 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Complex Post-Traumatic Stress Disorder
Keywords: mindfullness; treatment; compassion; trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TMC - group 1: TMC - group 1 was a closed group treated at a specialized outpatient facility for adult clients with CPTSD and complex dissociative disorders. Group 1 was led by two clinical psychologists
  Interventions: Other: TMC Treatment Approach
- TMC - group 2: TMC - group 2 was connected to specialized mental health services, but the intervention itself was carried out at a community centre. The community centre has collaborated with the District Psychiatric Centre (DPS) for many years, hosting an TMC group open to anyone attending the community centre in addition to clients connected to the DPS. This open concept was continued through the study intervention, but only clients connected to the DPS were included in the study.
  Interventions: Other: TMC Treatment Approach

INTERVENTIONS:
Other: TMC Treatment Approach — The TMC approach consists of 16 weekly group sessions, each lasting 2 hours. The first 10 sessions focus mainly on building mindfulness capacities, and the last 6 sessions on developing compassion toward self and others. Between sessions, participants are encouraged to do exercises with the support of audio files. The approach was developed with a transdiagnostic perspective, including clients with a variety of trauma-related symptoms.

SUMMARY:
This mixed-methods pilot study aim to assess the changes in symptoms of post-traumatic stress disorder (PTSD), complex post-traumatic stress disorder (CPTSD), dissociative symptoms, self-critique, and self-compassion following participation in a 16-week trauma-sensitive mindfulness and compassion (TMC) intervention. Adverse experiences of participation are also explored explicitly.

DETAILED DESCRIPTION:
Seventeen clients most female with severe childhood abuse and PTSD and CPTSD participated in the TMC intervention. A mixed-methods design was used. All clients completed questionnaires before (pre) and after (post) the intervention to gain information on symptom change, self-critique, and self-compassion. Second, a qualitative interview addressing clients' experiences of participation, including an explicit focus on adverse experiences, was conducted.

ELIGIBILITY:
Inclusion Criteria:

* report traumatic experiences and trauma related symptoms
* be between 18 and 65 years of age
* give informed consent to participate in the study

Exclusion Criteria:

* acute suicidality
* serious psychotic symptoms
* substance abuse interfering with treatment
* crisis interfering with treatment
* violent behavior

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion criteria in each group were in accordance with the institution's clinical practice
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for Diagnostic Statistical Manual (DSM) -5 | Change from pre-treatment to immediately after the intervention
  The Posttraumatic checklist (PCL-5) is a measure of perceived PTSD symptom severity in the past month. It was used to assess the likelihood of a PTSD diagnosis given 20 symptom descriptions (items) reflecting the DSM-5 criteria. Clients rated the extent to which they were troubled by PTSD symptoms on a 5-point Likert-type scale (0 for "Not at all" to 4 for "Extremely").

SECONDARY OUTCOMES:
The International Trauma Questionnaire (ITQ) | Change from pre-treatment to immediately after the intervention
  A 17-item self-report measure of ICD-11 PTSD and CPTSD were used to assess the CPTSD symptoms. Clients rated the extent to which they were troubled by CPTSD symptoms in the previous one month period on a 5-point Likert-type scale (0 for "Not at all to 4 for "Extremely"), reflecting the three clusters of disturbances in self-organization (DSO) in CPTSD (affective dysregulation, negative self-concept, and disturbances in relationships).
Trauma-Related Altered States of Consciousness (TRASC): | Change from pre-treatment to immediately after the intervention
  A 10-item self-report measure was used to survey a spectrum of dissociative experiences. Clients rated the extent to which they were troubled by TRASC symptoms on a 5-point Likert-type scale (0 for "Not at all" to 4 for "Extremely"). A total score was calculated across the items 1, 3, 5, 6, and 10 . Two items assessed depersonalization and derealization as in the Dissociative-PTSD subtype and the other items assessed the phenomenology of TRASC more broadly in reference to the subjective dimensions of time, thought, body, and emotion as per the 4-D model of trauma-related dissociation
General Anxiety Disorder-7 (GAD-7) | Change from pre-treatment to immediately after the intervention
  This symptom assessment tool measures anxiety with seven items in GAD-7 on a 4-point scale that assesses the impact on daily life.
Patient Health Questionnaire-9 (PHQ 9) | Change from pre-treatment to immediately after the intervention
  This symptom assessment tool measures depression with nine items in PHQ-9 on a 4-point scale that assesses the impact on daily life.
Self-Compassion Scale (SCS) | Change from pre-treatment to immediately after the intervention
  The 26-item SCS consists of three positive subscales, namely Self-Kindness (5 items), Common Humanity (4 items), and Mindfulness (4 items) and three negative subscales, namely Self-Judgment (5 items), Isolation (4 items), and Over-Identification (4 items). Respondents rate their agreement with items on a 5-point Likert-type scale from "Almost always" (5) to "Almost never" (1).

CONTACTS AND LOCATIONS:
Locations (1):
- Modum Bad, Vikersund, Norway

IPD SHARING:
Plan to Share IPD: Yes
The ethical approval granted by the Regional Committees for Medical and Health Research Ethics in Norway (REK and NSD) and in accordance with the information given to the participants in the informed consent form regarding the use of data, does not allow the authors to submit the data to a public repository. In line with the ethics approval, the data are to be kept at a secure server only accessible by the authors of this study. Access to the data can be granted following ethical approval of suggested project plan for the use of data from Modum Bad. The data will then be anonymized and further stored at a secure system. Such requests are to be sent to research leader, KariAnne Vrabel, Modum Bad, email: karianne.vrabel@modum-bad.no.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: It is already available at a secure server at modum bad. Hopefully, it will be published within next fall, 2023
Access Criteria: Placing the results of studies in a broader context: (for example, meta-analysis) Using the data as a convenience sample to address issues different from our research objectives Collaborating directly with other researchers where data need to be transferred to an alternative location for planned analyses connection of individual outcomes